CLINICAL TRIAL: NCT04505293
Title: Assessment of Accuracy, Precision, and Feasibility of a Handheld Near-Infrared Light Device (InfraScanner 2000™) in Detecting Subdural and Epidural Hematomas in Patients Admitted to Duke University Hospital and Mbarara Regional Referral Hospital: A Pilot Study
Brief Title: Assessment of InfraScanner 2000™ in Detecting Subdural and Epidural Hematomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00087011_1
Record Dates: First submitted 2020-07-22; First posted 2020-08-10 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Head Trauma; Craniocerebral Injuries; Crushing Skull Injury; Head Injuries; Head Injuries, Multiple; Head Injuries, Closed; Head Trauma,Closed; Head Trauma Injury; Head Trauma, Penetrating; Head Injury, Minor; Head Injury Major; Head Injury, Open; Injuries, Craniocerebral; Injuries, Head; Multiple Head Injury; Trauma, Head
MeSH Terms: conditions — Craniocerebral Trauma; Head Injuries, Closed; Head Injuries, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- InfraScanner 2000™ (Experimental): All patients entered onto the trial will undergo at least one cranial scanning using the InfraScanner 2000™ upon arrival to the casualty unit at MRRH following CT. Patients will be scanned using the InfraScanner 2000™ following each subsequent CT as allowed by patient or representative. Patients will know the results of the CT but not the InfraScanner 2000™. The standard for comparison will be determined as follows. A CT result that is positive for hematoma will be considered a true positive and a CT result that is negative for hematoma will be considered a true negative. In cases where the results of the CT are negative for hematoma and the results of the InfraScanner 2000™ are positive consideration of further follow-up will be given on a case-by-case basis.
  Interventions: Device: InfraScanner 2000™

INTERVENTIONS:
Device: InfraScanner 2000™ — The Infrascanner is a portable screening device that uses Near-Infrared (NIR) technology to screen patients for intracranial bleeding, identifying those who would most benefit from immediate referral to a CT scan and neurosurgical intervention.

SUMMARY:
The goal of this study is to determine the sensitivity, specificity, and positive and negative predictive values of the a portable near-infrared-based device (portable NIR-based device), the InfraScanner 2000™, to detect intracranial hematomas (epidural hematomas (EDH) and/or subdural hematomas (SDH)) in patients hospitalized at Mbarara Regional Referral Hospital (MRRH) who have sustained or who are suspected to have sustained head trauma.

DETAILED DESCRIPTION:
When applicable (conscious patient and/or family or legally authorized representative is present) the study will be introduced to the patient and relevant parties prior to the research team approaching the patient. While head trauma frequently results in impaired cognition and/or consciousness, and due to the urgency of these circumstances patients are often not accompanied by kin, whenever appropriate, the purpose of the research and the procedure will be explained in detail with all questions answered to the patient's and/or representative's satisfaction. Because patients who sustain head trauma injuries typically remain within the hospital for multiple days for monitoring and care, each participant may undergo multiple Computed Tomography (CT) scans over the course of his or her hospitalization, affording the opportunity of one to numerous measurements from each patient during his or her hospital stay.

Upon presentation to the casualty unit at MRRH and following each CT scan, the study team will approach the patient to scan the patient's cranium with the InfraScanner 2000™ (Image A). If permission is granted, the study team member sequentially measure the optical absorption for each of the 8 quadrants of the scalp (frontal, temporal, parietal, and occipital bilaterally) (Image B). The device is engineered such that the light emitter and receiver are spaced 4 cm apart, allowing the light's intensity to be measured between adjacent light guides (Image C). This entire procedure, including greeting and scanning the patient should take <10 minutes. Subsequent CT scan(s) the patient receives determines the number of potential data collections.

The patient and/or representative may refuse a scan during any encounter, and as such, the scan will not be done. For each patient scanned with the InfraScanner 2000™ they will be de-identified with a subject number, with age, sex, gender, skin color, hair color, hair thickness, mechanism of injury, Glasgow Coma Scale score, and mean time elapsed between CT scan and near-infrared measurement. These data will be stored in de-identified form on the Research Electronic Data Capture (REDCap) database and/or Microsoft Excel 2016 on a secured network drive within the Department of Neurosurgery at Duke.

The collection period for each research subject concludes 30-days following his or her initial measurement with the InfraScanner 2000™, patient discharge, or patient death.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who presents to MRRH with suspected head trauma, who is able to or who has a legally authorized representative who is able consent in English, Swahili, or Luganda will be considered for this study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haglund, MD, PhD, Principal Investigator — Duke University
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liow YY, Ukachukwu AK, Iversen ES, Ordonez YT, Gramer R, Shlobin NA, Najjuma JN, Fuller AT, Haglund MM, Kitya D, Kolls BJ. Assessment of a Handheld Near-Infrared Light Device in Detecting Intracranial Hematomas in Mbarara, Uganda. Neurosurgery. 2025 Dec 8. doi: 10.1227/neu.0000000000003873. Online ahead of print. PMID 41358727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mbarara Regional Referral Hospital in Mbarara, Uganda from the casualty ward. Participants were eligible for participation if they had a traumatic brain injury and could complete a CT and infrascan within 30 minutes of each other.
Period: Overall Study
Arm/Group | InfraScanner 2000™
Started | 672
Completed | 387
Not Completed | 285
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — CT scan unreadable | 277

BASELINE CHARACTERISTICS:
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 672
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.98 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 593
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 672
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 672
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Uganda | 672

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detection of Hematoma Stratified by CT Positive and CT Negative Status
Description: Determine whether the InfraScanner 2000 detects epidural and/or subdural hematomas with adequate precision relative to CT scans. Precision is defined as the number of True Positives (Infrascanner says there is a hematoma and the CT shows a hematoma) and True Negatives (Infrascanner says there is NOT a hematoma and the CT does NOT show a hematoma).
Time Frame: Within 30 minutes following CT scan
Population: 180 participants had a positive CT scan; 207 participants had a negative CT scan. One CT per participant.
Measure: Count of Participants; unit: Participants
Groups:
- InfraScanner 2000™ and CT (Computerized Tomography) Scan: All patients entered onto the trial will undergo at least one cranial scanning using the InfraScanner 2000™ upon arrival to the casualty unit at MRRH following CT. Patients will be scanned using the InfraScanner 2000™ following each subsequent CT as allowed by patient or representative. Patients will know the results of the CT but not the InfraScanner 2000™. The standard for comparison will be determined as follows. A CT result that is positive for hematoma will be considered a true positive and a CT result that is negative for hematoma will be considered a true negative. In cases where the results of the CT are negative for hematoma and the results of the InfraScanner 2000™ are positive consideration of further follow-up will be given on a case-by-case basis.
  InfraScanner 2000™: The Infrascanner is a portable screening device that uses Near-Infrared (NIR) technology to screen patients for intracranial bleeding, identifying those who would most benefit from immediate referral to a CT scan and neurosurgical intervention.
Arm/Group | InfraScanner 2000™ and CT (Computerized Tomography) Scan
Number analyzed (Participants) | 387
Participants
  CT positive: number analyzed (Participants) | 180
  CT positive: Infrascan positive | 158
  CT positive: Infrascan negative | 22
  CT negative: number analyzed (Participants) | 207
  CT negative: Infrascan positive | 126
  CT negative: Infrascan negative | 81

2. Secondary Outcome: Number of Participants With Detection of Hematoma Stratified by CT Positive and CT Negative Status (Adjusted for Volume and Size of Hematoma)
Description: Test characteristics of the InfraScanner 2000™ in identification of hematomas within its detection limits (volume >3.5 mL) compared to CT scan results as the gold standard. All CTs were reviewed to determine the size and depth from the skull of any hematomas present on the CT. All CT findings were used for the general analysis results to determine the number of True Positives and True Negatives. For the adjusted analyses (size and depth), only the CTs with hematoma sizes (>3.5 ml in volume) or depths (<2.5 cm from the skull) were used.
Time Frame: Within 30 minutes following CT scan
Population: Participants with hematomas within the InfraScanner's detection limits (as determined by CT scan). 151 participants had a positive CT scan and 207 participants had a negative CT scan when adjusted for hematoma volume/size. One CT per participant.
Measure: Count of Participants; unit: Participants
Arm/Group | InfraScanner 2000™ and CT (Computerized Tomography) Scan
Number analyzed (Participants) | 358
Participants
  CT positive (adjusted for volume/size): number analyzed (Participants) | 151
  CT positive (adjusted for volume/size): InfraScan positive (adjusted for volume/size) | 136
  CT positive (adjusted for volume/size): InfraScan negative (adjusted for volume/size) | 15
  CT negative (adjusted for size): number analyzed (Participants) | 207
  CT negative (adjusted for size): InfraScan positive (adjusted for volume/size) | 126
  CT negative (adjusted for size): InfraScan negative (adjusted for volume/size) | 81

3. Secondary Outcome: Number of Participants With Detection of Hematoma Stratified by CT Positive and CT Negative Status (Adjusted for Depth of Hematoma)
Description: Test characteristics of the InfraScanner 2000™ in identification of hematomas within its detection limits (depth <2.5 cm) compared to CT scan results as the gold standard. All CTs were reviewed to determine the size and depth from the skull of any hematomas present on the CT. All CT findings were used for the general analysis results to determine the number of True Positives and True Negatives. For the adjusted analyses (size and depth), only the CTs with hematoma sizes (>3.5 ml in volume) or depths (<2.5 cm from the skull) were used.
Time Frame: Within 30 minutes following CT scan
Population: Participants with hematomas within the InfraScanner's detection limits (as determined by CT scan). 165 participants had a positive CT scan and 207 participants had a negative CT scan when adjusted for hematoma depth. One CT per participant.
Measure: Count of Participants; unit: Participants
Arm/Group | InfraScanner 2000™ and CT (Computerized Tomography) Scan
Number analyzed (Participants) | 372
Participants
  CT positive (adjusted for depth): number analyzed (Participants) | 165
  CT positive (adjusted for depth): InfraScan positive (adjusted for depth) | 148
  CT positive (adjusted for depth): InfraScan negative (adjusted for depth) | 17
  CT negative (adjusted for depth): number analyzed (Participants) | 207
  CT negative (adjusted for depth): InfraScan positive (adjusted for depth) | 126
  CT negative (adjusted for depth): InfraScan negative (adjusted for depth) | 81

4. Secondary Outcome: Clinical Patient Outcomes as Measured by the Glasgow Outcomes Scale (GOSE)
Description: Clinical patient outcomes as measured by the Glasgow Outcomes Scale (GOSE) at discharge. The GOSE is rated from 1 to 8, 1 being death and 8 being upper good recovery.
Time Frame: Through study completion, defined as 30 days after CT scan or at discharge from hospital, death, or prior to leaving hospital against medical advice, whichever occurred first. All participants were assessed at a maximum of 30 days after CT scan.
Population: Data not collected on 10 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 377
Participants
  8 = Upper Good Recovery | 47
  7 = Lower Good Recovery | 252
  6 = Upper Moderate Disability | 41
  5 = Lower Moderate Disability | 9
  4 = Upper Severe Disability | 2
  3 = Lower Severe Disability | 0
  2 = Vegetative State | 0
  1 = Dead | 26

5. Secondary Outcome: Identify Reasons CT Not Performed
Description: CT Scans that are ordered and not performed will have a medical record review to determine the reasons for the missed CT.
Time Frame: as for outcome 4
Population: All CTs were performed.
Arm/Group | InfraScanner 2000™ and CT (Computerized Tomography) Scan
Number analyzed (Participants) | 0

6. Secondary Outcome: Causes of Head Trauma as Identified Through the Medical Record
Description: RTA = Road Traffic Accident
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 387
Participants
  RTA - Boda without helmet | 179
  RTA - Boda with helmet | 36
  RTA - Pedestrian hit by boda | 24
  RTA - Pedestrian hit by car or bus | 14
  RTA - Car without seatbelt | 12
  RTA - Car unknown seatbelt | 9
  RTA - Other | 17
  RTA - Car with seatbelt | 4
  RTA - Boda unknown helmet | 3
  Assault | 66
  Fall | 11
  Other | 6
  Accidental Injury | 4
  Unknown | 2

ADVERSE EVENTS:
Time Frame: Through study completion, defined as 30 days after CT scan or at discharge from hospital, death, or prior to leaving hospital against medical advice, whichever occurred first. All participants were assessed at a maximum of 30 days after CT scan.
Description: All-cause mortality instances were due to the participants' TBIs (traumatic brain injuries). Serious Adverse Events and/or Other (Not Including Serious) Adverse Events were not collected.
Arm/Group | InfraScanner 2000™ and CT (Computerized Tomography) Scan
All-Cause Mortality (participants affected / at risk) | 33/672
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04505293/Prot_SAP_000.pdf